CLINICAL TRIAL: NCT00358280
Title: A Randomised, Double-Blind, Multi-Centre, Parallel Group Study Comparing Efficacy and Safety of 5 mg/ml Ropivacaine and 5 mg/ml Bupivacaine for Spinal Anaesthesia in Patients Undergoing Unilateral Lower Limb Surgery
Brief Title: Ropivacaine Versus Bupivacaine for Spinal Anaesthesia in Patients Undergoing Unilateral Lower Limb Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D0695L00002
Record Dates: First submitted 2006-07-28; First posted 2006-07-31 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Anesthesia,Spinal
Keywords: Patients ASA category I ～ II; Unilateral Lower limb surgery; Spinal Anesthesia
MeSH Terms: interventions — Ropivacaine; Bupivacaine

INTERVENTIONS:
Drug: Ropivacaine
Drug: Bupivacaine

SUMMARY:
The purpose of this study is to compare the efficacy, duration of motor block until return to normal function in the non-operated leg after the start of injection, of ropivacaine 5 mg/ml and bupivacaine 5 mg/ml when used for spinal anaesthesia in patients undergoing unilateral lower limb surgery.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Men or women, 18 years £ age £ 70 years
* Patient scheduled for unilateral lower limb surgery with an estimated duration < 2 hours under spinal anaesthesia
* ASA category I ~ II
* 18.5 ≤ BMI ≤ 23.9

Exclusion Criteria:

* Contraindications to spinal anaesthesia, such as local infections, generalised septicaemia, platelet and clotting factor abnormalities, significant neurological disease with motor or sensory deficit, diagnosed increased intracranial pressure
* A known history of allergy, sensitivity or any other form of reaction to local anaesthetics of amide type
* Suspected inability to comply with the study procedures, including language difficulties or medical history and/or concomitant disease, as judged by the investigator
* Psychiatric history or any other concomitant disease which may lead to unreliability in clinical assessments, as judged by the investigator
* Significant alcohol, drug or medication abuse, as judged by the investigator
* Women who are pregnant or lactating or women of child bearing potential who are not practising adequate contraception or have positive urine pregnancy test (a urine Human chorionic gonadotropin [HCG] analysis)
* Involvement in the planning and conduct of the study (applies to both AstraZeneca staff or staff at the study site)
* Previous enrolment in the present study
* Participation in a clinical study during the last 3 months
* Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subjects' safety or successful participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2006-04; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy, duration of motor block until return to normal function in the non-operated leg after the start of injection, of ropivacaine 5 mg/ml and bupivacaine 5 mg/ml when used for spinal anaesthesia in patients undergoing unilateral lower

SECONDARY OUTCOMES:
To compare the efficacy of ropivacaine 5 mg/ml and bupivacaine 5 mg/ml in the duration of sensory block at dermatome T10 level
To compare the efficacy of ropivacaine 5 mg/ml and bupivacaine 5 mg/ml in the onset time of sensory block and motor block respectively
To compare the efficacy of ropivacaine 5 mg/ml and bupivacaine 5 mg/ml in the quality of anaesthesia
To compare the efficacy of ropivacaine 5 mg/ml and bupivacaine 5 mg/ml in subject pain during surgery
To determine the safety of ropivacaine 5 mg/ml and bupivacaine 5 mg/ml by evaluating the incidence and severity of adverse events, blood pressure, pulse rate and blood loss

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca China Medical Director, MD, Study Director — AstraZeneca
Locations (5):
- China (5):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Xi'an